CLINICAL TRIAL: NCT06658145
Title: The Establishment and Clinical Study of the Whole Visual VNOTES Approach Platform
Brief Title: Safety and Efficacy of Using a Novel Full Visual Access Platform System in Transvaginal Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jing Liang, Director of Obstetrics and Gynecology, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTCS-vnotesLH
Record Dates: First submitted 2024-09-10; First posted 2024-10-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-10

CONDITIONS: Uterine Myoma; Surgery, Laparoscopic
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full visibility vnotes group (Experimental): A suitable size of multi-channel vaginal sealing instrument was inserted from the vagina, pneumoperitoneum formed air pressure, and the vaginal dome was dilated and fully exposed. The dome was opened under laparoscopy, and an approach platform was established to complete the total hysterectomy.
  Interventions: Device: Vnotes surgery using fully visualised surgical instruments
- Traditional vnotes group (Experimental): The vaginal fornix and part of cervical ligaments were incised by vaginal operation, and an approach platform was established to complete hysterectomy.
  Interventions: Device: Vnotes surgery using traditional surgical instruments

INTERVENTIONS:
Device: Vnotes surgery using fully visualised surgical instruments — Vnotes surgery using fully visualised surgical instruments
  Arms: Full visibility vnotes group
Device: Vnotes surgery using traditional surgical instruments — Vnotes surgery using traditional surgical instruments
  Arms: Traditional vnotes group

SUMMARY:
The modified vNOTES hysterectomy was accomplished and validated for efficacy and safety using a multi-access vaginal confinement instrument with a fully visualised vaginal access platform.

DETAILED DESCRIPTION:
A multi-center prospective randomized controlled trial was conducted to evaluate the efficacy and safety of the vNOTES technique in patients with uterine fibroids who were scheduled for total hysterectomy. The patients were randomly assigned to the vNOTES group (experimental group) and the traditional vNOTES group (control group). The access platform was established using a visualization method or the traditional laparoscopic method, and the surgical operation was completed. The time required to establish the platform, the amount of bleeding, the total surgical time, the anesthesia indicators, complications, and follow-up indicators were recorded, and the effectiveness and safety of the technique were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≤ 60years old
2. Patients requiring total hysterectomy (with or without bilateral adjuncts or salpingectomy) due to uterine fibroids
3. BMI ranges from 18.5 to 27.9kg/m2;
4. Informed consent signed by the subject himself or his legal representative.

Exclusion Criteria:

1. Pregnant and lactating women;
2. asexual life history, vaginal malformations or adhesions, postmenopausal vaginal atrophy and stenosis;
3. Preoperative examination for malignant possibility
4. Uterine volume ≥20 weeks, history of pelvic inflammatory disease, severe endometriosis, degree III or IV uterine prolapse; Previous surgical history of intestinal obstruction, recurrent pelvic inflammatory disease, pelvic tuberculosis, and pelvic abdominal tumor; Gynecological examination of the uterine and rectal fossa is completely closed;
5. Patients known to have severe hepatic or renal dysfunction;
6. Patients with known blood disorders, coagulation disorders, active bleeding at any site, or bleeding propensity;
7. complicated with serious diseases of central nervous system, cardiovascular system, liver and kidney, digestive tract, respiratory system, endocrine and metabolism (thyroid disease, Cushing's syndrome, hyperprolactinemia), skeletal and muscular system and mental disorders;
8. patients with acute infection;
9. Known to have participated in any other clinical trial or taken hormone therapy within 3 months;
10. who cannot sign the informed consent;
11. For those with known or suspected poor compliance who could not complete the trial.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Success rate of access platform establishment | End of surgery
  Success is defined as opening the vaginal vault and entering the abdominal cavity to create stable abdominal pressure

SECONDARY OUTCOMES:
Tightness of equipment | End of surgery
  Throughout the operation, whether the device can remain airtight
Stability of equipment | End of surgery
  Throughout the operation, whether the equipment is tilted or slipped
Controllability of equipment | End of surgery
  Throughout the operation, whether the equipment can be smoothly inserted, extended, conformed, and advanced
Time of establishment of the access platform | End of surgery
  The time from the start of the procedure to the establishment of vaginal access
Total time of surgery | End of surgery
  The time from the beginning of the procedure to its complete completion
Total surgical bleeding volume | End of surgery
  Total blood loss from the beginning to the end of the procedure
The amount of bleeding during the process of establishing the platform | End of surgery
  The amount of bleeding from the beginning of surgery until the establishment of vaginal access
Surgical complications | 6 months after surgery
  Whether there was fever, infection and organ damage after operation
Length of hospital stay | 6 months after surgery
  The time from admission to discharge
Pain VAS score | 6 months after surgery
  Pain scores during postoperative hospital stay and follow-up（The Visual Analogue Scale (VAS) is a widely used method for pain assessment. 0 represents "no pain" and 10 represents "most severe pain".）
The Patients' life quality postoperative | 6 months after surgery
  The Patients' life quality postoperative be measured by Questionnaire.
Heart rate during surgery | End of surgery
  The magnitude of the change in the surgical center rate
blood pressure during surgery | End of surgery
  The magnitude of the change in blood pressure during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liang, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China